CLINICAL TRIAL: NCT00956683
Title: A Randomized Controlled Study Comparing Dual Endpoint Nerve Stimulation With Ultrasound-guided Infraclavicular Block for Hand Surgery.
Brief Title: Dual Endpoint Nerve Stimulation Versus Ultrasound in Infraclavicular Block for Hand Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Dr. Colin McCartney, University Health Network
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004-006
Record Dates: First submitted 2009-07-17; First posted 2009-08-11 (Estimated); Last update posted 2009-08-11 (Estimated); Status verified 2009-08

CONDITIONS: Hand Surgery
Keywords: infraclavicular nerve block ultrasound dual endpoint stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound (Experimental): Ultrasound guided infraclavicular block
  Interventions: Procedure: Ultrasound Guided Infraclavicular Nerve Block
- Dual Endpoint Nerve Stimulator (Active Comparator): Nerve stimulator guided dual endpoint infraclavicular block
  Interventions: Procedure: Dual-Endpoint nerve stimulation

INTERVENTIONS:
Procedure: Ultrasound Guided Infraclavicular Nerve Block — Use of Ultrasound to help guide needle placement and local anesthetic injection during infraclavicular nerve block.
  Arms: Ultrasound
Procedure: Dual-Endpoint nerve stimulation — Use of dual-endpoint nerve stimulation to guide needle placement and local anesthetic injection during infraclavicular nerve block.
  Arms: Dual Endpoint Nerve Stimulator

SUMMARY:
Current best practice for performance of infraclavicular block dictates the use of a dual-endpoint nerve stimulation technique that still only results in a 79% success rate. Use of an ultrasound-guided technique has the potential to significantly improve success. A randomized, controlled study to evaluate this area remains to be performed and is required to demonstrate to anesthesiologists that an ultrasound-guided approach should supersede nerve stimulation as the technique of choice for infraclavicular block.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective upper limb surgery at or below the elbow.
* Patients aged >18 and <80 years
* ASA I-III
* BMI<35

Exclusion Criteria:

* Inability to read, write or speak English. (This is necessary because subjects will have to follow detailed instructions to allow testing of motor and sensory function. It is not feasible to have an interpreter present in the block room during performance of these procedures)
* Contraindication to brachial plexus block
* Existing neurological deficit in the area to be blocked
* Known loco-regional malignancy or infection
* Coagulopathy
* Allergy to local anesthetic agents.
* Chest or shoulder deformities
* Severe respiratory disease
* Healed but dislocated clavicle fracture

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2006-01; Primary Completion 2008-08 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To compare ultrasound-guided infraclavicular block with conventional dual-endpoint nerve stimulator guided infraclavicular block with regards to block success, ease of nerve localization, speed of onset, duration of block and complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Colin McCartney, Toronto, Ontario, Canada